CLINICAL TRIAL: NCT05136885
Title: HEALEY ALS Platform Trial - Regimen E SLS-005 - Trehalose
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Seelos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518E
Record Dates: First submitted 2021-11-14; First posted 2021-11-29 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Regimen Specific Appendix; Lou Gehrig's Disease; Trehalose; Seelos Therapeutics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SLS-005 (Experimental): SLS-005 is administered via infusion once weekly for 24 weeks.
  Interventions: Drug: SLS-005
- Matching Placebo (Placebo Comparator): Matching placebo is administered via infusion once weekly for 24 weeks.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: SLS-005 — Administration: Infusion Dose: 0.75 g/kg weekly
  Arms: SLS-005
Drug: Matching Placebo — Administration: Infusion Dose: equivalent weight-based volume as described for trehalose
  Arms: Matching Placebo

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

Regimen E will evaluate the safety and efficacy of a single study drug, SLS-005 (Trehalose injection, 90.5 mg/mL for intravenous infusion) in participants with ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The HEALEY ALS Platform Trial Master Protocol is registered as NCT04297683.

Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

If a participant is randomized to Regimen E SLS-005 - Trehalose, the participant will complete a screening visit to assess additional Regimen E eligibility criteria. Once Regimen E eligibility criteria are confirmed, participants will complete a baseline assessment and be randomized in a 3:1 ratio to either active SLS-005 or matching placebo.

Regimen E will enroll by invitation, as participants may not choose to enroll in Regimen E. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen E.

For a list of enrolling sites, please see the HEALEY ALS Platform Trial Master Protocol under NCT04297683.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT NCT04297683).

Exclusion Criteria:

* The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT NCT04297683).

  1. Current diagnosis or healthcare professional-recommended treatment (medication, exercise or diet) of diabetes mellitus
  2. Master Protocol screening glucose >140 mg/dl
  3. Prior treatment with IV trehalose or known hypersensitivity to trehalose
  4. Current use of oral trehalose (see prohibited medication Section 5.9)
  5. Inability for participant to return to site for weekly drug administration, until approved for home infusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Healey Center for ALS at Mass General, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] HEALEY ALS Platform Trial; HEALEY ALS Platform Trial Study Group. Safety and efficacy of trehalose in amyotrophic lateral sclerosis (HEALEY ALS Platform Trial): an adaptive, phase 2/3, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2025 Jun;24(6):500-511. doi: 10.1016/S1474-4422(25)00173-5. PMID 40409314

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SLS-005 | Matching Placebo
Started | 120 | 41
Completed | 92 | 37
Not Completed | 28 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes only placebo participants from the Regimen E Efficacy Regimen Only (ERO) sample; shared placebo participants from other regimens are not included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | SLS-005 | Matching Placebo | Total
Number analyzed (Participants) | 120 | 41 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.73) | 61.3 (10.19) | 59.8 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 24 | 79
  Male | 65 | 17 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 115 | 40 | 155
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 109 | 39 | 148
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 3
ALS Diagnosis from R El Escorial Criteria [Count of Participants; unit: Participants] — The El Escorial Criteria are a set of guidelines used to diagnose ALS based on clinical signs of upper motor neuron and lower motor neuron dysfunction.
  Participants
    Clinically Definite ALS | 44 | 17 | 61
    Clinically Possible ALS | 8 | 3 | 11
    Clinically Probable ALS | 40 | 13 | 53
    Clinically Probable ALS - Laboratory Supported | 28 | 8 | 36
ALS Onset Location [Count of Participants; unit: Participants]
  Bulbar | 25 | 11 | 36
  Limb | 93 | 27 | 120
  Multiple | 2 | 1 | 3
  Respiratory | 0 | 2 | 2
Time Since Symptom Onset at Baseline [Mean (Standard Deviation); unit: Months] | 19.6 (8.61) | 19.9 (8.20) | 19.7 (8.48)
Delay in ALS Symptom Onset and Diagnosis [Mean (Standard Deviation); unit: Months] | 10.7 (6.86) | 10.1 (4.82) | 10.5 (6.39)
Baseline Edaravone Use [Count of Participants; unit: Participants]
  No | 84 | 28 | 112
  Yes | 36 | 13 | 49
Baseline Riluzole Use [Count of Participants; unit: Participants]
  No | 33 | 11 | 44
  Yes | 87 | 30 | 117
ALSFRS-R Total Score [Mean (Standard Deviation); unit: Points] — The ALS Functional Rating Score-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
  Points | 35.8 (6.43) | 35.0 (6.71) | 35.6 (6.49)
Baseline Decline in ALSFRS-R [Mean (Standard Deviation); unit: points per month] — The ALS Functional Rating Score-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function. Baseline is divided by the number of months between onset of weakness due to ALS and the date of Baseline. A higher number indicates greater decline.
  points per month | 0.76 (0.608) | 0.76 (0.504) | 0.76 (0.582)
SVC [Mean (Standard Deviation); unit: percent predicted] — Slow vital capacity is an assessment of breathing function. The total amount of air that can be exhaled is measured. A higher slow vital capacity indicates better breathing function. Population: Number analyzed in row differs from overall number due to missing data.
  percent predicted
    number analyzed (Participants) | 119 | 41 | 160
    (all) | 74.5 (18.81) | 77.9 (16.54) | 75.4 (18.26)
King Stage [Count of Participants; unit: Participants] — The King's ALS Clinical Staging System is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction. Level 4a indicates nutritional failure and level 4b indicates respiratory failure. Higher scores indicate a worse disease state.
  Participants
    1 Region with Neuromuscular Dysfunction | 20 | 8 | 28
    2 Region with Neuromuscular Dysfunction | 38 | 13 | 51
    3 Region with Neuromuscular Dysfunction | 36 | 5 | 41
    4a/b Nutritional/Respiratory Failure | 26 | 15 | 41
Weight [Mean (Standard Deviation); unit: kg] | 79.3 (21.44) | 76.8 (17.65) | 78.6 (20.52)
Body Mass Index [Mean (Standard Deviation); unit: kg/cm^2] | 26.7 (6.47) | 26.8 (5.15) | 26.7 (6.14)
Serum Creatinine Concentration [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.19) | 0.7 (0.16) | 0.7 (0.18)
Serum NfL Concentration [Mean (Standard Deviation); unit: ng/L] — Population: Number analyzed in row differs from overall number due to missing data.
  ng/L
    number analyzed (Participants) | 116 | 39 | 155
    (all) | 76.9 (51.08) | 76.5 (38.45) | 76.8 (48.09)

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Assessed by the ALSFRS-R Slope
Description: Change in disease severity over time as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R). Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
Time Frame: 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set, which included shared placebo from other regimens, as pre-specified in the Regimen Statistical Analysis Plan. Regimen A (NCT04436497), Regimen B (NCT04436510), Regimen C (NCT04414345) and Regimen D (NCT04615923) contributed placebo participants into the shared placebo cohort used for analysis.
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | SLS-005 | Matching Placebo
Number analyzed (Participants) | 120 | 204
points per month | -0.91 (0.090) | -1.06 (0.091)
Statistical Analysis 1: Comparison: SLS-005 vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter model — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. (Trehalose) slowed progression) was (0.8772). NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 0.87, 95% CI 2-sided [0.665 to 1.102], Standard Deviation 0.111 — DDR <1 imply slowing of disease progression by Trehalose relative to placebo.Note: reported "Confidence Interval" is actually a Bayesian credible interval; The DRR parameter for active treatment represents the relative change to the rate of decline of ALSFRS-R and the rate of mortality of treated participant relative to a placebo participant. The estimated DRR can also be interpreted as the average rate of decline in function and mortality. The model includes covariates for baseline use of edaravone, baseline use of riluzole, baseline use of Relyvrio, months since onset of symptoms, and pre-baseline slope of ALSFRS-R, serum NfL concentration and random effects for regimen and participant-specific slopes

2. Primary Outcome: Mortality Event Rate
Description: Mortality is defined as death or death equivalent. A participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row. The rate of mortality was estimated from a Bayesian shared-parametric model that assumed exponentially distributed survival times.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per month
Arm/Group | SLS-005 | Matching Placebo
Number analyzed (Participants) | 120 | 204
events per month | 0.010 (0.0025) | 0.012 (0.0027)

3. Secondary Outcome: Respiratory Function
Description: Change in respiratory function over time as measured by Slow Vital Capacity (SVC).
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set, which included shared placebo from other regimens, as pre-specified in the Regimen Statistical Analysis Plan. Regimen A (NCT04436497), Regimen B (NCT04436510), Regimen C (NCT04414345) and Regimen D (NCT04615923) contributed placebo participants into the shared placebo cohort used for analysis.One SLS-005 participant and 4 placebo participants from FAS were not analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | SLS-005 | Matching Placebo
Number analyzed (Participants) | 119 | 201
percent change | -11.40 (1.431) | -10.85 (1.089)
Statistical Analysis 1: Comparison: SLS-005 vs Matching Placebo; Test type: Superiority; p = 0.7607, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, pre-baseline ALSFRS-R slope, and baseline log-transformed NfL; Mean Difference (Net) = -0.55, 95% CI 2-sided [-4.06 to 2.97], Standard Error of Mean 1.790 — Trehalose 24-week change from baseline relative to placebo 24-week change from baseline

4. Secondary Outcome: Muscle Strength
Description: Change in muscle strength over time as measured isometrically using hand-held dynamometry (HHD).
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set, which included shared placebo from other regimens, as pre-specified in the Regimen Statistical Analysis Plan. Regimen A (NCT04436497), Regimen B (NCT04436510), Regimen C (NCT04414345) and Regimen D (NCT04615923) contributed placebo participants into the shared placebo cohort used for analysis. Two placebo participants from FAS were not analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | SLS-005 | Matching Placebo
Number analyzed (Participants) | 120 | 203
percent change | -26.19 (2.568) | -27.11 (1.876)
Statistical Analysis 1: Comparison: SLS-005 vs Matching Placebo; Test type: Superiority; p = 0.7737, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = 0.92, 95% CI 2-sided [-5.37 to 7.21], Standard Error of Mean 3.204 — Trehalose 24-week change from baseline relative to placebo 24-week change from baseline

5. Secondary Outcome: Number of Participants That Experienced Death or Death Equivalent
Description: The number of participants who died or met the criterion for a death equivalent from the date of their baseline visit to the end of the Week 24 visit window (generally 175 days after baseline). The death equivalent criterion is the use of permanent assisted ventilation (PAV) for more than 22 hours per day for more than 7 days in a row.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SLS-005 | Matching Placebo
Number analyzed (Participants) | 120 | 203
Participants | 10 | 10
Statistical Analysis 1: Comparison: SLS-005 vs Matching Placebo; Test type: Superiority; p = 0.2137, Log Rank

ADVERSE EVENTS:
Time Frame: Up to 35 weeks after participant signed Master Protocol consent.
Arm/Group | SLS-005 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 6/120 | 0/41
Serious Adverse Events (participants affected / at risk) | 19/120 | 3/41
Other Adverse Events (participants affected / at risk) | 107/120 | 33/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLS-005 (N=120) | Matching Placebo (N=41)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Urticaria (Immune system disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLS-005 (N=120) | Matching Placebo (N=41)
Muscular weakness (Nervous system disorders) | 22 (30) | 8 (14)
Neuromyopathy (Nervous system disorders) | 18 (22) | 4 (5)
Headache (Nervous system disorders) | 11 (15) | 0 (0)
Dysarthria (Nervous system disorders) | 4 (4) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 32 (63) | 8 (17)
Infusion site bruising (Injury, poisoning and procedural complications) | 7 (12) | 2 (2)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 8 (10) | 0 (0)
Fatigue (General disorders) | 19 (20) | 6 (7)
Infusion related reaction (General disorders) | 6 (33) | 2 (30)
Oedema peripheral (General disorders) | 6 (7) | 2 (4)
Constipation (Gastrointestinal disorders) | 15 (16) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (15) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 9 (10) | 2 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 4 (4) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 0 (0)
COVID-19 (Infections and infestations) | 12 (12) | 3 (3)
Urinary tract infection (Infections and infestations) | 7 (10) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT05136885/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT05136885/SAP_001.pdf